CLINICAL TRIAL: NCT02164071
Title: Validation of a Comprehensive Health Status Assessment Scale in Elderly Patients (≥ 65 Years) With Hematological Malignancies
Acronym: GAH
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: CEL-GAH-2011-01
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Myelodysplastic Syndromes; Leukemia Myeloid Acute; Multiple Myeloma; Leuklemia, Lymphocytic, Chronic
Keywords: Haematological malignancy; Elderly; Health Status; Scale validation
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Multiple Myeloma; Bronchiolitis Obliterans Syndrome; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Multiple Myeloma (MM): Patients with Myltiple Myeloma, symptomatic or asymptomatic
  Interventions: Other: Geriatric Assessment of Health Status Scale administration
- Myelodysplastic Syndromes or Acute Myeloid Leukemia: Patients with Myelodysplastic Syndromes (MDS), any International Prognostic Scoring System (IPSS) risk, or Acute Myeloid Leukemia (AML)
  Interventions: Other: Geriatric Assessment of Health Status Scale administration
- Chronic Lymphocytic Leukemia (CLL): Patients with Chronic Lymphocytic Leukemia
  Interventions: Other: Geriatric Assessment of Health Status Scale administration

INTERVENTIONS:
Other: Geriatric Assessment of Health Status Scale administration — Scale will be administered to all patients (3 cohorts) at baseline and then after 5 and not more than 15 days
  Other Names: Geriatric Assessment of Health Status Scale

SUMMARY:
The elderly comprise the most prevalent population in oncology practice. The available evidence suggests that old patients are undertreated patients, mainly because of their advanced age, regardless of whether they are highly functional patients, they do not present co morbidities and could benefit from oncology therapies.

Treatment planning must consider several health indices that are useful when it comes to detecting geriatric problems that could affect the patient's treatment experience. The complete comprehensive geriatric evaluation stands out as cornerstone among other validated tools that do not work as isolated instruments; however, its length and complexity may hinder its routine use in clinical practice for decision making.

The purpose of this study is to validate a comprehensive health status assessment scale in elderly patients (≥65 years) with hematological malignancies that, while integrating the essential dimensions of geriatric assessment and, with the same precision as the currently available valid tools, is shorter and easier to apply, so it can be incorporated into the daily practice and that aids in clinical decision making objectively.

If so, this information would help identify patients that could benefit from a specific oncology treatment, thus contributing to developing a targeted intervention plan and to optimizing the cancer results in this patient population.

ELIGIBILITY:
Inclusion Criteria:

Patients ≥ 65 years old. Treatment-naïve patients

Newly diagnosed patients who belong to one of the 3 following groups:

Patients with MDS (any risk grade as per IPSS) or AML Patients with multiple myeloma (symptomatic or not) or Patients with chronic lymphocytic leukemia (including A status) Patients who have granted their informed consent.

Exclusion Criteria:

Not fulfilling selection criteria

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Eligible patients, even being naïve to treatment, are eligible to receive treatment at any time as per clinical practice. Patients ≥ 65 years old, newly diagnosed, naïve to treatment, belonging to one of the 3 following groups. 1.- Patients with Myelodysplastic Syndromes (any risk according to) or Acute myeloid leukemia; 2.- Patients with Multiple Myeloma, either symptomatic or asymptomatic; or 3.- Patients with Chronic lymphocytic leukemia (including stadium A).
Sampling Method: Non-Probability Sample
Enrollment: 363 (Actual)
Dates: Start 2012-04-11 (Actual); Primary Completion 2013-12-03 (Actual); Study Completion 2015-07-04 (Actual)

PRIMARY OUTCOMES:
Geriatric Health Assessment (GHA) Questionnaire | Approximately 2.5 years
  A composite variable comprised of all the dimensions that make up the GHA questionnaire will be obtained on stable patients as a result of the implementation of a questionnaire by two independent evaluators: one investigator and one duly trained health professional.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Luis Garcia, PhD, Study Director — Celgene
Locations (22):
- Spain (22):
  - Hospital Txagorritxu, Vitoria-Gasteiz, Alava
  - Hospital Sant Joan de Deu, Espluges de Llobregat, Barcelona
  - Hospital Duran I Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital Parc Tauli, Sabadell, Barcelona
  - Hospital de Donostia, Donostia / San Sebastian, Guipuzcoa
  - Hospital U. Puerta de Hierro, Majadahonda, Madrid
  - C.H. Navarra, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Hospital Ntra. Sra. La Candelaria, Santa Cruz de Tenerife, Tenerife
  - Hospital La Ribera, Alzira, Valencia
  - C.H. Universitario A Coruna, A Coruña
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clinic, Barcelona
  - Hospital Virgen de las Nieves, Granada
  - Arnau de Vilanova, Lleida
  - Hospital U. Gregorio Maranon, Madrid
  - Hospital Infanta Leonor, Madrid
  - Hospital de Segovia, Segovia
  - Hospital Virgen del Rocio, Seville
  - Hospital La Fe, Valencia